CLINICAL TRIAL: NCT04826276
Title: Effects of Smoking State on Effort-based Decision Making
Brief Title: Effects of Smoking State on Decision Making
Acronym: Effort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00079949
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2022-09

CONDITIONS: Behavior
Keywords: Decision making
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be instructed to smoke as usual before one fMRI study visit (satiated state) and to abstain from using all tobacco/nicotine for 12 hours before the other fMRI study visit (abstinence and/or withdrawn state). The order of the satiated and abstinence/withdrawn study visits will be randomized and counterbalanced across participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Subjects (Experimental): for the abstinence intervention, 12+ hours after smoking will be assessed before assessments following smoking as normal
  For the satiated intervention, smoking as normal will be assessed first before assessments following 12+ hours of abstinence from smoking
  Interventions: Other: smoking abstinence; Other: smoking satiety

INTERVENTIONS:
Other: smoking abstinence — participants will be asked to not smoke for at least 12 hours
Other: smoking satiety — participants will be asked to smoke as usual

SUMMARY:
Adult smokers will be tested using behavioral and neuroimaging measures after smoking as usual and after overnight abstinence.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-55 years
* Smokes cigarettes or e-cigarettes
* Negative urine drug screen

Exclusion Criteria:

* Unstable or serious medical or mental health condition
* History of serious head trauma
* Pregnancy
* Unsuitable for MRI
* Weight > 350 pounds (maximum allowed for MRI)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Effort based decision making | through study completion, an average of 1 year
  number of high effort selections
Distress tolerance behavior | through study completion, an average of 1 year
  duration on measures of distress tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Merideth Addicott, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT04826276/ICF_000.pdf